CLINICAL TRIAL: NCT02075931
Title: Collaborative-care Intervention to Promote Physical Activity After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-2568
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Feedback (Experimental): The physical activity feedback intervention will involve real-time physical activity monitoring using a device to provide activity feedback directly to patients in combination with patient group meetings held monthly during the 12 week intervention for the purposes of mutual support in attaining physical activity goals.
  Interventions: Other: Physical activity feedback with group meetings
- Control (Active Comparator): The control represents the current standard of care post total knee arthroplasty.
  Interventions: Other: Control

INTERVENTIONS:
Other: Physical activity feedback with group meetings — Physical activity feedback
  Arms: Physical Activity Feedback
Other: Control — No intervention
  Arms: Control

SUMMARY:
The investigators have learned that knee replacement patients are not more physically active after surgery. This is true even though their pain is less compared to before surgery. This low level of physical activity is not healthy. It can increase the chances of weight gain, which can create other issues. It can also lessen physical function. Some studies have looked at physical activity feedback systems to increase how active people are. Studies have investigated face to face patient group meetings for this,too. These systems and meetings can increase physical activity. The investigators will study the effects of a physical activity monitors with group meetings after knee replacement. The investigators hypothesize that physical activity levels and physical function will increase. The investigators goal is to help knee replacement patients lead healthier lives and maintain or enhance their physical function.

DETAILED DESCRIPTION:
More than 650,000 total knee arthroplasties (TKAs) are performed annually to alleviate pain and disability associated with osteoarthritis (OA); a chronic, degenerative condition that compromises the quality of life of 37% of adults over age 60. With the aging of the population, an estimated 3.5 million TKAs will be performed annually by 2030. Despite improvements in pain and self-reported function, physical activity after TKA remains at pre-operative, sedentary levels (<5,000 steps/day). Physical activity in TKA confers powerful protective effects against common post-surgical sequelae including increased weight gain (mean=6.4 kg, 2 years post TKA), decreased functional performance, increased risk/progression of co-morbid conditions (e.g. type 2 diabetes mellitus, cardiovascular disease), and progression of knee and hip osteoarthritis which may necessitate additional joint replacement in the contralateral limb. An intervention aimed at improved self-management of physical activity may aid patients in overcoming habitual lifestyle patterns of low physical activity secondary to knee pain prior to TKA.

Recent investigations on the effects of real-time, user-friendly, electronic physical activity feedback (PAF) systems and face-to-face (FTF) patient group meetings aimed to promote self-management of physical activity suggest that such interventions can successfully increase physical activity. Therefore, the investigators propose a randomized, controlled trial to assess efficacy and feasibility of a physical activity intervention combined with FTF group meetings (PAF+FTF) initiated within one month of patients' discharge from outpatient rehabilitation for TKA compared to a control group receiving standard care (CON). This type of intervention is surprisingly novel to this patient population and is not common practice in rehabilitation following TKA.

ELIGIBILITY:
Inclusion Criteria:

* undergone unilateral total knee arthroplasty

Exclusion Criteria:

* severe contralateral leg osteoarthritis (>4/10 with stair climbing)
* unstable orthopaedic condition that limits function
* neurological conditions that affect muscle function
* vascular or cardiac conditions that limit function

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity | Change from baseline to immediately post-12 week intervention
  Daily step and activity counts

SECONDARY OUTCOMES:
Change in Functional performance | Change from baseline to immediately post-12 week intervention
  Six-minute walk test, timed up-and-go, 10 meter walk test
Change in Self-reported physical function | Change from baseline to immediately post-12 week intervention
  Knee injury and Osteoarthritis Outcome Score, Physical Activity Scale for the Elderly

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens-Lapsley, MPT, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States